CLINICAL TRIAL: NCT01170221
Title: A Phase 3 Randomized, Double-Blind, Multicenter Study Comparing the Efficacy and Safety of 6-Day Oral TR-701 Free Acid and 10-Day Oral Linezolid for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Brief Title: TR-701 FA vs. Linezolid for the Treatment of Acute Bacterial Skin and Skin Structure Infections.
Acronym: ABSSSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1986-009; TR701-112 (Other: TriusRX Unique ID)
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Skin and Subcutaneous Tissue Bacterial Infections
Keywords: ABSSSI; Tedizolid Phosphate; TR-701; Acute Bacterial Skin and Skin Structure Infections
MeSH Terms: interventions — tedizolid phosphate; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TR-701 FA (Experimental): TR0-701 FA 200 mg tablets once a day for six days followed by 4 days of placebo
  Interventions: Drug: TR-701 FA
- Linezolid (Active Comparator): Linezolid 600 mg tablets oral twice a day for 10 days
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: TR-701 FA — Oral TR-701 FA 200 mg once daily for six days followed by four days of placebo.
  Other Names: Tedizolid Phosphate; TR-700 active moiety
  Arms: TR-701 FA
Drug: Linezolid — Oral Linezolid 600 mg twice daily for 10 days
  Other Names: Trade name = Zyvox; Generic name = linezolid
  Arms: Linezolid

SUMMARY:
This is a randomized, double-blind, double dummy, multicenter Phase 3 study of oral TR-701 FA 200 mg once daily for 6 days versus oral Zyvox® (linezolid) 600 mg every 12 hours for 10 days for the treatment of ABSSSI in adults.

Approximately 75 to 100 sites globally will participate in this study. Patients with an ABSSSI caused by suspected or documented gram positive pathogen(s) at baseline will be randomized 1:1 to study treatment

DETAILED DESCRIPTION:
The primary objective is to determine the noninferiority in the early clinical response rate of 6 day oral TR-701 FA compared with that of 10-day oral linezolid treatment at the 48-72 Hour Visit in the ITT analysis set in patients with ABSSSI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic signs of infection diagnosed with acute bacterial skin and skin structure infection (ABSSSI)
* Diagnosed with Cellulitis/ erysipelas, major cutaneous abscess, or wound infections

Exclusion Criteria:

* Uncomplicated skin infections
* Severe sepsis or septic shock
* ABSSSI solely due to gram-negative pathogens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2010-08-15 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Prokocimer, MD, Study Director — Trius Therapeutics
Locations (84):
- United States (30):
  - Trius investigator site 109, Dothan, Alabama
  - Trius Investigator site 130, Anaheim, California
  - Trius investigator site 118, Anaheim, California
  - Trius investigator site 129, Buena Park, California
  - Trius Investigator Site 103, Chula Vista, California
  - Trius Investigator Site 105, La Mesa, California
  - Trius investigator site 126, Laguna Beach, California
  - Trius investigator site 125, Norwalk, California
  - Trius Investigator Site 104, Oceanside, California
  - Trius investigator site 113, Oxnard, California
  - Trius investigator site 123, Pasadena, California
  - Trius Investigator Site 106, Rolling Hills Estates, California
  - Trius investigator site 111, Torrance, California
  - Trius investigator site 132, Torrance, California
  - Trius investigator site 127, Fort Lauderdale, Florida
  - Trius investigator site 135, Hialeah, Florida
  - Trius investigator site 101, Columbus, Georgia
  - Trius Investigator Site 102, Savannah, Georgia
  - Trius Investigator site 116, Chicago, Illinois
  - Trius Investigator Site 108, Springfield, Illinois
  - Trius investigator site 112, Evansville, Indiana
  - Trius Investigator Site 107, Detroit, Michigan
  - Trius investigator site 133, Butte, Montana
  - Trius investigator site 128, Las Vegas, Nevada
  - Trius investigator site 115, Somers Point, New Jersey
  - Trius investigator site 114, Toledo, Ohio
  - Trius investigator site 122, Houston, Texas
  - Trius investigator site 120, Houston, Texas
  - Trius investigator site 131, Houston, Texas
  - Trius Investigator site 121, Houston, Texas
- Argentina (10):
  - Trius investigator site 307, Avellaneda, Pcia Buenos Aires
  - Trius investigator site 304, Loma Hermosa, Pcia Buenos Aires
  - Trius investigator site 309, Buenos Aires
  - Trius investigator site 310, Buenos Aires
  - Trius Investigator site 301, Córdoba
  - Trius investigator site 305, Córdoba
  - Trius investigator site 300, Córdoba
  - Trius investigator site 308, Paraná
  - Trius investigator site 303, Rosario
  - Trius investigator site 306, Santa Fe
- Brazil (4):
  - Trius investigator site 322, Barro Preto, Belo Horizonte
  - Trius investigator site 321, São José do Rio Preto, São Paulo
  - Trius investigator site 323, São Paulo, São Paulo
  - Trius investigator site 320, Belo Horizonte
- Canada (6):
  - Trius investigator site 170, Winnipeg, Manitoba
  - Trius investigator site 172, Hamilton, Ontario
  - Trius investigator site 171, Hamilton, Ontario
  - Trius investigator site 175, Brownsburg, Quebec
  - Trius investigator site 173, Chicoutimi, Quebec
  - Trius investigator site 174, Sherbrooke, Quebec
- Czechia (5):
  - Trius investigator site 234, Hradec Králové
  - Trius investigator site 235, Mělník
  - Trius investigator site 233, Ostrava
  - Trius investigator site 236, Pardubice
  - Trius investigator site 231, Prague
- Germany (4):
  - Trius investigator site 201, Berlin
  - Trius investigator site 202, Hanau
  - Trius investigator site 200, Mannheim
  - Trius investigator site 203, Plauen
- Hungary (3):
  - Trius investigator site 241, Debrecen
  - Trius investigator site 242, Komló
  - Trius investigator site 240, Szeged
- Latvia (4):
  - Trius investigator site 258, Daugavpils
  - Trius investigator site 256, Liepāja
  - Trius investigator site 257, Rēzekne
  - Trius investigator site 255, Riga
- Peru (4):
  - Trius investigator site 343, Lima Cercado, Lima region
  - Trius investigator site 342, Miraflores, Lima region
  - Trius investigator site 341, San Juan de Miraflores, Lima region
  - Trius investigator site 340, Arequipa
- Slovakia (2):
  - Trius investigator site 251, Banská Bystrica
  - Trius investigator site 250, Martin
- Ukraine (12):
  - Trius investigator site 271, Cherkassy
  - Trius investigator site 264, Dnipro
  - Trius investigator site 263, Dnipro
  - Trius investigator site 269, Ivano-Frankivsk
  - Trius investigator site 260, Kharkiv
  - Trius investigator site 261, Kyiv
  - Trius investigator site 268, Lviv
  - Trius investigator site 265, Lviv
  - Trius Investigator site 270, Ternopil
  - Trius investigator site 266, Uzhhorod
  - Trius investigator site 262, Zaporizhzhya
  - Trius investigator site 267, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Sandison T, De Anda C, Fang E, Das AF, Prokocimer P. Clinical Response of Tedizolid versus Linezolid in Acute Bacterial Skin and Skin Structure Infections by Severity Measure Using a Pooled Analysis from Two Phase 3 Double-Blind Trials. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e02687-16. doi: 10.1128/AAC.02687-16. Print 2017 May. PMID 28264845
- [Derived] Nathwani D, Corey R, Das AF, Sandison T, De Anda C, Prokocimer P. Early Clinical Response as a Predictor of Late Treatment Success in Patients With Acute Bacterial Skin and Skin Structure Infections: Retrospective Analysis of 2 Randomized Controlled Trials. Clin Infect Dis. 2017 Jan 15;64(2):214-217. doi: 10.1093/cid/ciw750. Epub 2016 Dec 21. PMID 28003218
- [Derived] Powers JH 3rd, Das AF, De Anda C, Prokocimer P. Clinician-reported lesion measurements in skin infection trials: Definitions, reliability, and association with patient-reported pain. Contemp Clin Trials. 2016 Sep;50:265-72. doi: 10.1016/j.cct.2016.08.010. Epub 2016 Aug 13. PMID 27530088
- [Derived] Shorr AF, Lodise TP, Corey GR, De Anda C, Fang E, Das AF, Prokocimer P. Analysis of the phase 3 ESTABLISH trials of tedizolid versus linezolid in acute bacterial skin and skin structure infections. Antimicrob Agents Chemother. 2015 Feb;59(2):864-71. doi: 10.1128/AAC.03688-14. Epub 2014 Nov 24. PMID 25421472
- [Derived] Lodise TP, Fang E, Minassian SL, Prokocimer PG. Platelet profile in patients with acute bacterial skin and skin structure infections receiving tedizolid or linezolid: findings from the Phase 3 ESTABLISH clinical trials. Antimicrob Agents Chemother. 2014 Dec;58(12):7198-204. doi: 10.1128/AAC.03509-14. Epub 2014 Sep 22. PMID 25246392
- [Derived] Bien P, De Anda C, Prokocimer P. Comparison of digital planimetry and ruler technique to measure ABSSSI lesion sizes in the ESTABLISH-1 study. Surg Infect (Larchmt). 2014 Apr;15(2):105-10. doi: 10.1089/sur.2013.070. Epub 2014 Jan 22. PMID 24450727
- [Derived] Prokocimer P, De Anda C, Fang E, Mehra P, Das A. Tedizolid phosphate vs linezolid for treatment of acute bacterial skin and skin structure infections: the ESTABLISH-1 randomized trial. JAMA. 2013 Feb 13;309(6):559-69. doi: 10.1001/jama.2013.241. PMID 23403680

RESULTS

PARTICIPANT FLOW:
Groups:
- Tedizolid Phosphate: Oral Tedizolid phosphate 200 mg once daily for six days followed by four days of placebo
Period: Overall Study
Arm/Group | Tedizolid Phosphate | Linezolid
Started | 332 | 335
Completed | 299 | 307
Not Completed | 33 | 28
Not completed — Lost to Follow-up | 22 | 21
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Subject completed only screening and LFU | 1 | 0
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Tedizolid Phosphate | Linezolid | Total
Number analyzed (Participants) | 332 | 335 | 667
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (14.96) | 43.1 (15.06) | 43.3 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 137 | 265
  Male | 204 | 198 | 402

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response Rate
Description: Responder: No increase in lesion surface area from baseline and oral temperature ≤37.6°C
Time Frame: 48-72 hours
Population: The ITT analysis set includes data from all randomized participants.
Measure: Number; unit: Responders
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 335
Responders | 264 [-6.1 to 6.2] | 266 [-6.1 to 6.2]
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; The primary objective is to determine the noninferiority in the early clinical response rate of oral tedizolid phosphate compared with that of oral linezolid treatment at the 48-72 Hour Visit in the ITT Analysis Set in patients with ABSSSI; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI for the observed difference in the primary outcome measure (early clinical response at the 48-72 Hour Visit) between the tedizolid group and the linezolid group was calculated using the ITT analysis set. Noninferiority was concluded if the lower limit of the 95% CI was greater than -10%; Risk Difference (RD) = 0.1, 95% CI [-6.1 to 6.2] — Risk difference corresponds to tedizolid clinical response rate minus linezolid clinical response rate. The confidence interval was calculated using the Miettinen and Nurminen with stratification for the presence or absence of fever at baseline

2. Secondary Outcome: Clinical Response at 48-72 Hours That is Sustained at the End of Therapy Visit.
Description: Responder: No increase in lesion surface area from baseline and oral temperature ≤37.6°C.
Time Frame: Day 11
Population: The ITT analysis set includes data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 335
participants | 230 | 241
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI will be calculated for the observed differences in the clinical response rate based on the sustained response at EOT using the method of Miettinen and Nurminen with stratification for the presence or absence of fever at baseline. Noninferiority was concluded if the lower limit of the 95% CI was greater than -10% and the conditions of the hierarchical testing procedure were met; Hierarchical testing procedure of Westfall and Krishen used to control for inflation of the overall type I error rate. If NI is declared for the primary, NI will be tested for the secondary outcomes in this order: Secondary Outcomes Measures 2 to 5; Risk Difference (RD) = -2.6, 95% CI 2-sided [-9.6 to 4.2] — Risk difference corresponds to the tedizolid clinical response rate minus the linezolid clinical response rate

3. Secondary Outcome: Clinical Response at 48-72 Hours That is Sustained at the End of Therapy Visit in the Clinically Evaluable-End of Therapy Analysis Sets
Description: Responder: No increase in lesion surface area from baseline and oral temperature ≤37.6°C
Time Frame: EOT Day 11
Population: All randomized patients receiving minimal study therapy, completed 48-72 Hour and EOT assessments, no concomitant systemic antibiotic therapy through EOT, and had no confounding events or factors
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 273 | 286
participants | 219 | 232
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was calculated for the observed differences in the clinical response rate based on the sustained response at EOT using the method of Miettinen and Nurminen with stratification for the presence or absence of fever at baseline. Noninferiority was concluded if the lower limit of the 95% CI was greater than -10% and the conditions of the hierarchical testing procedure were met; Risk Difference (RD) = -0.9, 95% CI 2-sided [-7.7 to 5.4] — Risk difference corresponds to the tedizolid clinical response rate minus the linezolid clinical response rate

4. Secondary Outcome: Investigator's Assessment of Clinical Success at the Post Treatment Evaluation Visit
Description: Clinical success defined as resolution/near resolution of most disease-specific signs and symptoms, absence/near resolution of systemic signs of infection, if present at baseline, no new signs, symptoms, or complications attributable to the ABSSSIs so no further antibiotic therapy was required for the treatment of the primary lesion.
Time Frame: Post-Treatment Evaluation (7-14 days after the End of Therapy)
Population: The Intent to Treat analysis set included data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 335
participants | 284 | 288
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was calculated for the observed differences in the clinical success rate based on the Investigator's assessment of clinical response at the PTE visit using the method of Miettinen and Nurminen with stratification for the presence or absence of fever at baseline. Noninferiority was concluded if the lower limit of the 95% CI was greater than -10% and the conditions of the hierarchical testing procedure were met; Risk Difference (RD) = -0.5, 95% CI 2-sided [-5.8 to 4.9] — Risk difference corresponds to the tedizolid clinical success rate minus the linezolid clinical success rate

5. Secondary Outcome: To Compare the Investigator's Assessment of Clinical Success at the Post Treatment Evaluation Visit in the Clinically Evaluable-Post Treatment Evaluation Analysis Set
Description: Clinical success defined as resolution/near resolution of most disease-specific signs and symptoms, absence/near resolution of systemic signs of infection, no new signs, symptoms, or complications attributable to the ABSSSIs so no further antibiotic therapy was required for the treatment of the primary lesion.
Time Frame: Post-Treatment Evaluation (7-14 days after the End of Therapy)
Population: All randomized patients who received the minimal study therapy, completed EOT and PTE assessments, no concomitant systemic antibiotic therapy through PTE, and had no confounding events or factors.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 279 | 280
participants | 264 | 267
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Risk Difference (RD) = -0.8, 95% CI 2-sided [-4.6 to 3.0] — Risk difference corresponds to the tedizolid clinical success rate minus the linezolid clinical success rate

6. Secondary Outcome: Investigator's Assessment of Clinical Response at the 48-72 Hour Visit
Description: Clinical improvement was defined as improvement in overall clinical status.
Time Frame: 48-72 Hour Visit
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 335
participants | 299 | 290
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; A two-sided 95% CI was calculated for the observed differences in the clinical response rate based on the Investigator's assessment of clinical response at the 48-72 Hour Visit using the method of Miettinen and Nurminen with stratification for the presence or absence of fever at baseline; Test type: Superiority or Other; Risk Difference (RD) = 3.5, 95% CI 2-sided [-1.4 to 8.5] — Risk difference corresponds to the tedizolid clinical response rate minus the linezolid clinical response rate

7. Secondary Outcome: Investigator's Assessment of Clinical Response at the Day 7 Visit
Description: Clinical improvement was defined as improvement in overall clinical status.
Time Frame: Day 7
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Number; unit: participants
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 335
participants | 302 | 299
Statistical Analysis 1: Comparison: Tedizolid Phosphate vs Linezolid; A two-sided 95% CI was calculated for the observed differences in the clinical response rate based on the Investigator's assessment of clinical response at the Day 7 Visit using the method of Miettinen and Nurminen with stratification for the presence or absence of fever at baseline; Test type: Superiority or Other; Risk Difference (RD) = 1.7, 95% CI 2-sided [-2.8 to 6.4] — Risk difference corresponds to the tedizolid clinical response rate minus the linezolid clinical response rate

8. Secondary Outcome: Change From Baseline in Patient-reported Pain, by Study Visit
Description: 0=no pain, 10=worst pain Only 1 visit per participant for Day 4-6, only 1 visit for Day 7-9, and only 1 visit for Day 10-13.
Time Frame: Multiple
Population: The Intent to Treat analysis set includes data from all randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tedizolid Phosphate | Linezolid
Number analyzed (Participants) | 332 | 335
units on a scale
  Day 2 | -1.3 (2.05) | -1.5 (1.99)
  Day 4-6 | -3.4 (2.44) | -3.1 (2.41)
  Day 7-9 | -4.5 (2.71) | -4.6 (2.67)
  Day 10-13 | -5.3 (2.65) | -5.5 (2.58)

ADVERSE EVENTS:
Time Frame: Collected from signing of the ICF through the late follow-up visit (up to 38 days).
Description: Numbers for at risk include all treated participants.
Arm/Group | Tedizolid Phosphate | Linezolid
Serious Adverse Events (participants affected / at risk) | 5/331 | 4/335
Other Adverse Events (participants affected / at risk) | 84/331 | 100/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tedizolid Phosphate (N=331) | Linezolid (N=335)
Cardiac arrest (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Alcoholic psychosis (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tedizolid Phosphate (N=331) | Linezolid (N=335)
Nausea (Gastrointestinal disorders) | 28 | 45
Headache (Nervous system disorders) | 21 | 17
Diarrhea (Gastrointestinal disorders) | 15 | 18
Abscess (Infections and infestations) | 14 | 8
Abscess limb (Infections and infestations) | 12 | 10
Vomiting (Gastrointestinal disorders) | 9 | 20
Cellulitis (Infections and infestations) | 8 | 8
Dizziness (Nervous system disorders) | 8 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 8
Dyspepsia (Gastrointestinal disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to pursue publication of results in cooperation with a lead Investigator, subject to the terms and conditions of the clinical study agreement between the Sponsor and Investigators. Sponsor approval is required for publication of any data subsets. Final authorship will be determined in accordance with the International Committee of Medical Journal Editors definition of authorship.